CLINICAL TRIAL: NCT02517788
Title: Comparative Pharmacokinetic Profile of Interferon Beta-1a (Bioferon®) Administered as Single i.v. Doses in HSA-free Formulation and HSA+ Solution and as Multiple s.c. Doses in Healthy Subjects
Brief Title: Phase I BP Interferon (IFN) Beta-004
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: BioPartners GmbH (Industry)
Responsible Party: Principal Investigator, Prof. Jérôme Biollaz, MD, Chief Physician, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CE 93/06; 2006DR1162 (Registry Identifier: Swissmedic)
Record Dates: First submitted 2015-08-05; First posted 2015-08-07 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-08

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Interferon beta-1a

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Part A: Interferon beta-1a in HSA-free solution (Experimental): Twelve subjects will participate in 3 periods of part A, receiving 18 MIU biosimilar interferon beta-1a without albumin as i.v. bolus into a distal port under constant saline infusion as 3 treatments.
  Interventions: Drug: Interferon beta-1a HSA-free biosimilar
- Part A: Interferon beta-1a combined with HSA+ solution (Experimental): Twelve subjects will participate in 3 periods of part A, receiving 18 MIU biosimilar interferon beta-1a with albumin as i.v. bolus into a distal port under constant saline infusion as 3 treatments.
  Interventions: Drug: Interferon beta-1a HSA+ biosimilar
- Part A: Interferon beta-1a in marketed HSA+ solution (Active Comparator): Twelve subjects will participate in 3 periods of part A, receiving 18 MIU original interferon beta-1a with albumin as i.v. bolus into a distal port under constant saline infusion as 3 treatments.
  Interventions: Drug: Interferon beta-1a original
- Part B: Interferon beta-1a in HSA-free solution (Experimental): Twelve additional volunteers will participate in part B, receiving 4 x 18 MIU biosimilar interferon beta-1a with albumin as s.c. doses at 48 hours intervals as 3 pre-filled syringes (3 sites 1 cm apart in abdominal wall on each dosing day, alternating right side for odd dose [i.e. dose 1 and 3] and left side for even dose [i.e. dose 2 and 4]).
  Interventions: Drug: Interferon beta-1a HSA-free biosimilar
- Part B: Interferon beta-1a in marketed HSA+ solution (Active Comparator): Part B: Twelve additional volunteers will participate in part B, receiving 4 x 18 MIU original interferon beta-1a with albumin as s.c. doses at 48 hours intervals as 3 pre-filled syringes (3 sites 1 cm apart in abdominal wall on each dosing day, alternating right side for odd dose [i.e. dose 1 and 3] and left side for even dose [i.e. dose 2 and 4]).
  Interventions: Drug: Interferon beta-1a original

INTERVENTIONS:
Drug: Interferon beta-1a HSA-free biosimilar — 6 MIU/0.53 mL in pre-filled glass syringe solubilized in aqueous isotonic buffered solution without albumin
  Other Names: Bioferon®
  Arms: Part A: Interferon beta-1a in HSA-free solution; Part B: Interferon beta-1a in HSA-free solution
Drug: Interferon beta-1a HSA+ biosimilar — 6 MIU/0.53 mL in pre-filled glass syringe solubilized in aqueous isotonic buffered solution combined with albumin solution
  Other Names: Bioferon®
  Arms: Part A: Interferon beta-1a combined with HSA+ solution
Drug: Interferon beta-1a original — 6 MIU/0.50 mL in pre-filled glass syringe solubilized in HSA and mannitol solution (marketed formulation)
  Other Names: Rebif®
  Arms: Part A: Interferon beta-1a in marketed HSA+ solution; Part B: Interferon beta-1a in marketed HSA+ solution

SUMMARY:
Phase I study aiming at:

* establishing the pharmacokinetic profile of interferon beta-1a after i.v. administration of the formulation BioPartners IFN beta-1a without albumin (HSA-free solution in pre-filled syringes) at 18 MIU;
* investigating the possible impact of albumin on pharmacokinetic profile by comparing 3 different i.v. formulations: BioPartners IFN beta-1a without albumin (HSA-free solution in pre-filled syringes), BioPartners IFN beta-1a with added albumin (HSA+), and Rebif® from Merck-Serono, a registered IFN beta-1a solution containing HSA;
* establishing the steady state pharmacokinetic profile of BioPartners IFN beta-1a in HSA-free solution after 4 subsequent s.c. doses of 18 MIU given at 48 hour intervals against Rebif® using the same regimen.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects aged between 18 and 45 years
* Weight range between 55 and 95 kg for males, 45 and 80 kg for females, providing body mass index (BMI) was between 18 and 29 kg/m2
* Absence of significant findings in the medical history and physical examination
* Absence of significant laboratory abnormalities as judged by the investigator.
* 12-lead ECG without significant abnormalities
* Negative urine drug screen

Exclusion Criteria:

* History of major renal, hepatic, immunological, haematological, gastrointestinal, genitourinary, neurological, or rheumatological disorders
* Active diseases of any type, even if mild, including inflammatory disorders and infections.
* Pregnant or lactating women or women contemplating becoming pregnant during study. Female subjects of child-bearing potential who did not practice efficient contraception during the study. A pregnancy test in blood was performed at screening and before each period with β-human chorionic gonadotropin for females of child-bearing potential. If pregnancy test was positive, the subject had to be immediately excluded from study and followed until delivery
* History of severe allergy or of asthma at any time.
* History of cardiovascular dysfunction
* Hypertension
* Sick sinus syndrome or known long QT syndrome
* Presence of QTc ￼ > 440 msec or pronounced sinus bradycardia (<40 bpm/min), even if elicited by sport
* Dark skin preventing local tolerance assessment or abnormal cutaneous reaction e.g. urticaria or papular dermographism
* Intense sport activities.
* Any clinically significant laboratory value on screening that were not within normal range on single repeat
* Positive hepatitis B & C antigen screen
* Positive HIV antibody screen or screen not performed
* Any recent acute illness or sequelae thereof which could expose the subject to a higher risk or might confound the results of the study
* Treatment in the previous three months with any drug known to have well-defined potential for toxicity to a major organ
* History of hypersensitivity to any drug if considered as serious
* History of alcohol or drug abuse
* Positive qualitative urine drug test at screening
* Use of any medication in 2 weeks prior to study and throughout study, including aspirin or other over-the-counter preparation.
* Blood (500 mL) donation or hemorrhage during the previous three months
* Participation in a clinical trial in the previous 3 months
* Smoking
* Consumption of a large quantity of coffee, tea or equivalent
* Present consumption of a large quantity of alcohol or wine or equivalent
* Psychological status which could have had an impact on subject's ability to give informed consent or behavioral tests
* Any feature of subject's medical history or present condition which, in the investigator's opinion, could confound the results of the study, complicate its interpretation, or represent a potential risk for the subject

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2006-05; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Composite of interferon beta-1a PK parameters | Part A: 0, 2, 5, 10, 15, 20 [min post-dose] and 0.5, 0.75, 1, 2, 3, 4, 6, 8, 12, 24 [hours post-dose] / Part B: 0, 1, 2, 3, 4, 6, 12 [hours post-doses] and 0, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168 [hours post-last dose] (Day 7)
  Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUC[0-inf]) and maximum observed concentration (Cmax) following single dose administration, as well as time to Cmax (tmax; for s.c. injection) will be assessed. Mean residence time (MRT), half-life of elimination (t1/2), clearance (CL), and volume of distribution at steady-state (Vss) will be calculated.

SECONDARY OUTCOMES:
Serum concentration of neopterin (PD marker) | Part A: 0, 6, 12, 24, 48, 72, 168 [hours post-doses] / Part B: 0, 6, 12 [hours post-doses] and 0, 6, 12, 24, 48, 72, 96, 120, 144, 168 [hours post-last dose] (Day 7)
  Assessment by ELISA after i.v. and after s.c
Number of participants with adverse events (AE)/serious adverse event (SAE) as a measure of safety and tolerability | Up to Day 7
  AE/SAE will be collected from the start of study treatment and until the follow-up visit
Composite of local reactions as a measure of local tolerance | Part A: 0, 0.5, 1, 2, 4, 6, 8, 10, 12, 24 [hours post-dose] and longer if needed and until resolution in case of local reaction / Part B: 0, 1, 2, 4, 6, 12 [hours post-dose] on Day 1 and 7, else daily up to Day 9 longer until resolution
  Any local symptoms rated as moderate (grade 3 for i.v. and 2 for s.c.) or severe (grade 4 and 5 for i.v.; grade 3 for s.c.) will be reported as an adverse event. The subjective painful sensation following injection of the drug will be assessed using a visual analogue scale (VAS)
Composite of clinical laboratory tests as a measure of safety and tolerability | Screening and 0, 24 [hours post-doses]
  Clinical laboratory tests will include hematology, clinical chemistry and urinalysis
Composite of vital signs as a measure of safety and tolerability | Part A: Screening and 0, 1, 2, 3, 4, 6, 8, 10, 12, 24 [hours post-dose] / Part B: Screening and 0, 1, 2, 3, 4, 6, 12 [hours post-doses], as well as 0, 1, 2, 3, 4, 6, 8, 12, 24 [hours post-last dose] (Day 7)
  Vital signs will include body temperature, blood pressure and heart rate
Sickness behavior assessment | Part A: 0, 2, 4, 6, 8, 10, 12 [hours post-dose] / Part B: 0, 1, 2, 4, 6, 12 [hours post-dose], as well as 24, 48, 72 [hours post-last dose] (Day 7)
  Four parameters will be recorded (general feeling, headache, muscle ache, mood)
Electrocardiogram (ECG) as a measure of safety and tolerability | Screening and 0, 3 [hours post-dose]
  Twelve-lead ECG will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme Biollaz, MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois

REFERENCES:
- [Derived] Perrottet N, Brunner-Ferber F, Grouzmann E, Spertini F, Biollaz J, Buclin T, Widmer N. Biases affecting injected doses of an experimental drug during clinical trials. Trials. 2016 Jul 16;17(1):321. doi: 10.1186/s13063-016-1463-5. PMID 27423899